CLINICAL TRIAL: NCT04595357
Title: "Iris Shelf" Technique for Intraocular Foreign Bodies Removal
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Abdelazeem, Associate professor of Ophthalmology, Assiut University
Other Study IDs: 17300500
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Eye Injuries
MeSH Terms: conditions — Eye Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Iris shelf technique — Removal of posterior segment intraocular foreign bodies through corneal incision combined with phaco-vitrectomy

SUMMARY:
Intraocular foreign body (IOFB) injury is a common potentially serious form of ocular trauma. Metallic IOFB is the most common type of IOFB injury. Apart from the associated ocular tissue damage, Metallic IOFB may cause permanent visual impairment due to retinal toxicity and endophthalmitis.

When presenting posteriorly, the approach of IOFB removal is challenging. Several techniques had been described for posterior IOFB removal. All of these techniques aimed to remove IOFB with the least possible collateral damage. This study aims to describe "Iris shelf" technique for posterior IOFB removal through a clear corneal incision combined with phaco-vitrectomy and report its outcomes.

ELIGIBILITY:
Inclusion Criteria:

- posterior segment metallic IOFB who underwent combined phacovitrectomy with IOFB removal through a clear corneal incision using "Iris shelf" technique

Exclusion Criteria:

* Any other surgical technique for posterior segment IOFB removal

Ages: 15 Years to 45 Years | Sex: All
Age Groups: Child, Adult
Study Population: patients with posterior segment metallic IOFB who underwent combined phacovitrectomy with IOFB removal through a clear corneal incision using "Iris shelf" technique at Assiut University hospitals and Al-Forsan eye center, Assiut; Egypt in the period between January 2016 and December 2019.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
corrected distance visual acuity | 1 month

IPD SHARING:
Plan to Share IPD: No